CLINICAL TRIAL: NCT00665769
Title: Physiological Disturbances Associated With Neonatal Intraventricular Hemorrhage
Acronym: PhysDis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was proceeding too slowly
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Christopher J. Rhee, MD, MS, Professor of Pediatrics and Obstetrics and Gynecology, Baylor University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-31475; 1R01NS060674 (NIH)
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Intraventricular Hemorrhage; Autoregulation
Keywords: hypercapnia; normocapnia; chronic lung disease; periventricular leukomalacia; intraventricular hemorrhage; hypotension; cerebral autoregulation; heart rate variability; autonomic nervous system; detrended fluctuation analysis
MeSH Terms: conditions — Hypercapnia; Leukomalacia, Periventricular; Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypercapnia (Placebo Comparator): Hypercapnic ventilation. The goal will be to maintain transcutaneous CO2 55 mm Hg (50-60 mm Hg) during the first week of life, or until extubation. A written, laminated hypercapnic ventilator algorithm will be placed at the bedside.
  Interventions: Other: Hypercapnia
- Normocapnia (Active Comparator): Normocapnic ventilation. The goal will be to maintain transcutaenous CO2 40 mm Hg (35-45 mm Hg) during the first week of life, or until extubation. A written, laminated normocapnic ventilator algorithm will be placed at the bedside.
  Interventions: Other: Normocapnia

INTERVENTIONS:
Other: Hypercapnia — transcutaenous CO2 50-60 mm Hg
  Other Names: hypercarbia; permissive hypercapnia
  Arms: Hypercapnia
Other: Normocapnia — transcutaneous CO2 35-45 mm Hg
  Other Names: Normocarbia
  Arms: Normocapnia

SUMMARY:
Annually, almost 5,000 extremely low birth weight (9 ounces to about 2 lbs) infants born in the US survive with severe bleeding in the brain (intraventricular hemorrhage); this devastating complication of prematurity is associated with many problems, including mental retardation, cerebral palsy, and learning disabilities, that result in profound individual and familial consequences. In addition, lifetime care costs for these severely affected infants born in a single year exceed $3 billion. The huge individual and societal costs underscore the need for developing care strategies that may limit severe bleeding in the brain of these tiny infants. The overall goal of our research is to evaluate disturbances of brain blood flow in these tiny infants in order to predict which of them are at highest risk and to develop better intensive care techniques that will limit severe brain injury.

1. Since most of these infants require ventilators (respirators) to survive, we will investigate how 2 different methods of ventilation affect brain injury. We believe that a new method of ventilation, allowing normal carbon dioxide levels, will normalize brain blood flow and lead to less bleeding in the brain.
2. We will also examine how treatment for low blood pressure in these infants may be associated with brain injury. We believe that most very premature infants with low blood pressure actually do worse if they are treated. We think that by allowing the infants to normalize blood pressure on their own will allow them to stabilize blood flow to the brain leading to less intraventricular hemorrhage.
3. In 10 premature infants with severe brain bleeding, we have developed a simple technique to identify intraventricular hemorrhage before it happens. Apparently, the heart rate of infants who eventually develop severe intraventricular hemorrhage is less variable than infants who do not develop this. We plan to test this method in a large group of infants, to be able to predict which infants are at highest risk of developing intraventricular hemorrhage and who could most benefit from interventions that would reduce disturbances of brain blood flow.

ELIGIBILITY:
Inclusion Criteria:

* ventilated ELBW (401-1000 grams) infants
* 23 to 30 weeks' gestation
* umbilical arterial catheter placed during newborn resuscitation

Exclusion Criteria:

* presence of complex congenital anomalies or chromosomal abnormality
* presence of central nervous system malformation
* infants with hydrops fetalis
* infants in extremis
* infants with early (<3 hour of age) intraventricular hemorrhage

Ages: 1 Minute to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2008-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The effect of hypercapnia vs. normocapnia on the development of Grade II-IV intraventricular hemorrhage/periventricular leukomalacia (severe brain injury) and/or death | During first 2 weeks of life (intraventricular hemorrhage and/or death), initial hospitalization for periventricular leukomalacia

SECONDARY OUTCOMES:
The effect of hypercapnia vs. normocapnia on the development of chronic lung disease (requirement of supplemental oxygen at 36 weeks corrected gestational age) | By 36 weeks corrected gestational age.
The effect of hypercapnia vs. normocapnia on abnormal results from MRIs | at term-equivalent age
The effect of hypercapnia vs. normocapnia on the development of pulmonary hemorrhage | During the initial hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R. Kaiser, MD, MA, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Background] Hall RW, Kaiser JR. Hypotension and brain injury in premature infants. Pediatrics. 2008 Mar;121(3):654; author reply 654-5. doi: 10.1542/peds.2007-3602. No abstract available. PMID 18310222
- [Background] Kaiser JR, Gauss CH, Williams DK. Tracheal suctioning is associated with prolonged disturbances of cerebral hemodynamics in very low birth weight infants. J Perinatol. 2008 Jan;28(1):34-41. doi: 10.1038/sj.jp.7211848. Epub 2007 Oct 25. PMID 18165829
- [Background] Kaiser JR. Both extremes of arterial carbon dioxide pressure and the magnitude of fluctuations in arterial carbon dioxide pressure are associated with severe intraventricular hemorrhage in preterm infants. Pediatrics. 2007 May;119(5):1039; author reply 1039-40. doi: 10.1542/peds.2007-0353. No abstract available. PMID 17473113
- [Background] Kaiser JR, Gauss CH, Pont MM, Williams DK. Hypercapnia during the first 3 days of life is associated with severe intraventricular hemorrhage in very low birth weight infants. J Perinatol. 2006 May;26(5):279-85. doi: 10.1038/sj.jp.7211492. PMID 16554847
- [Background] Kaiser JR, Gauss CH, Williams DK. The effects of hypercapnia on cerebral autoregulation in ventilated very low birth weight infants. Pediatr Res. 2005 Nov;58(5):931-5. doi: 10.1203/01.pdr.0000182180.80645.0c. PMID 16257928
- [Background] Kaiser JR, Gauss CH, Williams DK. Surfactant administration acutely affects cerebral and systemic hemodynamics and gas exchange in very-low-birth-weight infants. J Pediatr. 2004 Jun;144(6):809-14. doi: 10.1016/j.jpeds.2004.03.022. PMID 15192631
- [Background] Tuzcu V, Nas S, Borklu T, Ugur A. Decrease in the heart rate complexity prior to the onset of atrial fibrillation. Europace. 2006 Jun;8(6):398-402. doi: 10.1093/europace/eul031. Epub 2006 May 10. PMID 16687424
- [Background] Rushing S, Ment LR. Preterm birth: a cost benefit analysis. Semin Perinatol. 2004 Dec;28(6):444-50. doi: 10.1053/j.semperi.2004.10.007. PMID 15693401
- [Background] van Bel F, de Winter PJ, Wijnands HB, van de Bor M, Egberts J. Cerebral and aortic blood flow velocity patterns in preterm infants receiving prophylactic surfactant treatment. Acta Paediatr. 1992 Jun-Jul;81(6-7):504-10. doi: 10.1111/j.1651-2227.1992.tb12283.x. PMID 1392362
- [Background] van de Bor M, Walther FJ. Cerebral blood flow velocity regulation in preterm infants. Biol Neonate. 1991;59(6):329-35. doi: 10.1159/000243368. PMID 1873365
- [Background] Lou HC, Lassen NA, Friis-Hansen B. Impaired autoregulation of cerebral blood flow in the distressed newborn infant. J Pediatr. 1979 Jan;94(1):118-21. doi: 10.1016/s0022-3476(79)80373-x. PMID 758388
- [Background] Fabres J, Carlo WA, Phillips V, Howard G, Ambalavanan N. Both extremes of arterial carbon dioxide pressure and the magnitude of fluctuations in arterial carbon dioxide pressure are associated with severe intraventricular hemorrhage in preterm infants. Pediatrics. 2007 Feb;119(2):299-305. doi: 10.1542/peds.2006-2434. PMID 17272619
- [Background] Fanaroff JM, Wilson-Costello DE, Newman NS, Montpetite MM, Fanaroff AA. Treated hypotension is associated with neonatal morbidity and hearing loss in extremely low birth weight infants. Pediatrics. 2006 Apr;117(4):1131-5. doi: 10.1542/peds.2005-1230. PMID 16585307
- [Background] van Ravenswaaij-Arts CM, Hopman JC, Kollee LA, van Amen JP, Stoelinga GB, van Geijn HP. The influence of respiratory distress syndrome on heart rate variability in very preterm infants. Early Hum Dev. 1991 Dec;27(3):207-21. doi: 10.1016/0378-3782(91)90195-9. PMID 1802672